CLINICAL TRIAL: NCT03547154
Title: A RANDOMIZED PHASE 2/3 TRIAL OF SCH 54031 PEG12000 INTERFERON ALFA-2b (PEG INTRON, SCH 54031) VS. INTRON A (SCH 30500) IN SUBJECTS WITH NEWLY DIAGNOSED CML (PROTOCOL NOS. C/I98-026)
Brief Title: Polyethylene Glycol Interferon Alfa-2b (PEG Intron) Versus Interferon Alfa-2b (INTRON^® A) in the Treatment of Newly Diagnosed Chronic Myelogenous Leukemia (CML) (C98026)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C98026; MK-4031-001 (Other: Merck Protocol Number); C98-026 (Other: Schering-Plough)
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — peginterferon alfa-2b; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegylated interferon alfa-2b (Experimental): Participants received pegylated interferon alfa-2b (PEG Intron) at a dose of 6.0 microg/kg, administered weekly by subcutaneous (SC) injection. Participants may have received hydroxyurea therapy as needed prior to randomization to reduce or keep the white blood cell (WBC) count ≤50,000/μl. Treatment was for a minimum of 6 months unless there was evidence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pegylated interferon alfa-2b
- Interferon alfa-2b (Active Comparator): Participants received interferon alfa-2b (Intron^® A), recombinant for injection, at a dose of 5 million international units (MIU)/m^2, administered daily by SC injection. Participants may have received hydroxyurea therapy as needed prior to randomization to reduce or keep the WBC count ≤50,000/μl. Treatment was for a minimum of 6 months unless there was evidence of disease progression or unacceptable toxicity.
  Interventions: Biological: Interferon alfa-2b

INTERVENTIONS:
Biological: Pegylated interferon alfa-2b — Weekly SC injection of pegylated interferon alfa-2b, 6.0 microg/kg
  Other Names: PEG Intron
  Arms: Pegylated interferon alfa-2b
Biological: Interferon alfa-2b — Daily SC injection of interferon alfa-2b, 5 MIU/m^2
  Other Names: INTRON^® A
  Arms: Interferon alfa-2b

SUMMARY:
The primary purpose of this study is to compare the efficacy of polyethylene glycol (PEG; pegylated) interferon alfa-2b (PEG Intron, C98026) versus interferon alfa-2b (Intron® A) in the treatment of participants with newly diagnosed CML.

ELIGIBILITY:
Inclusion Criteria

* Has chronic phase CML diagnosed within 3 months prior to study enrollment
* Has chronic phase CML positive for Ph^1 as confirmed by cytogenetic studies, performed by a central laboratory
* Has platelet count >/= 50,000/microl
* Has hemoglobin >/= 9.0 g/dL
* Has WBC count >/=2000/microl but </= 50,000/microl
* Has adequate hepatic and renal function, as defined by the following parameters obtained within 14 days prior to initiation of study treatment

  * serum glutamic oxaloacetic transaminase (SGOT) <2 times upper limit of laboratory normal (ULN)
  * serum glutamic pyruvic transaminase SGPT <2 times upper ULN
  * serum bilirubin <2 times ULN
  * serum creatinine <2.0 mg/dL
* Is fully recovered from any prior major surgery and must be at least 4 weeks postoperative
* Has Eastern Cooperative Oncology Group Performance Status of 0-2
* Has signed a written, voluntary informed consent before study entry, is willing to participate in this study, and is willing to complete all follow-up assessments

Exclusion Criteria:

* Has accelerated phase CML as defined by any of the following criteria.

  * peripheral blood myeloblasts >/=15%
  * peripheral blood basophils >/= 20%
  * peripheral blood myeloblasts plus promyelocytes >/=30%
  * platelets <100,000/microl, unrelated to therapy
* Has blastic phase CML (30% myeloblasts in peripheral blood or bone marrow)
* Is a candidate for and is planning to receive allogeneic, syngeneic, or autologous bone marrow transplantation within the next 12 months
* Has received prior treatment for their CML, except for hydroxyurea (collection of stem cells without using high dose chemotherapy for mobilization is acceptable)
* Has severe cardiovascular disease (i. e., arrhythmias requiring chronic treatment, congestive heart failure [New York Heart Association (NYHA) Class III or IV], or symptomatic ischemic heart disease)
* Has a history of a neuropsychiatric disorder requiring hospitalization
* Has thyroid dysfunction not responsive to therapy
* Has uncontrolled diabetes mellitus
* Has a history of seropositivity for human immunodeficiency virus
* Has active and/or uncontrolled infection, including active hepatitis
* Has a medical condition requiring chronic systemic corticosteroids
* Has a history of prior malignancies within the last 5 years, except for surgically cured non-melanoma skin cancer, or cervical carcinoma in situ
* Has received any experimental therapy within 30 days prior to enrollment in this study
* Is known to be actively abusing alcohol or drugs
* Is pregnant, nursing, or of reproductive potential and is not practicing an effective means of contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 1998-10-22 (Actual); Primary Completion 2001-02-20 (Actual); Study Completion 2001-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- INTRON A (Interferon Alfa-2b): Interferon alfa-2b, recombinant for injection, 5 million international units (MIU)/m^2, administered daily by SC injection. Treatment was for a minimum of 6 months (mo.) unless there was evidence of disease progression or unacceptable toxicity.
- PEG Intron (Pegylated Interferon Alfa-2b): Pegylated interferon alfa-2b, 6.0 microg/kg, administered weekly by subcutaneous (SC) injection. Treatment was for a minimum of 6 months unless there was evidence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | INTRON A (Interferon Alfa-2b) | PEG Intron (Pegylated Interferon Alfa-2b)
Started | 173 | 171
Completed | 50 | 55
Not Completed | 123 | 116
Not completed — Disease Progression/Recurrence | 6 | 14
Not completed — Adverse Event | 26 | 31
Not completed — Protocol Violation | 6 | 1
Not completed — Physician Decision | 4 | 3
Not completed — Insufficient Therapeutic Response | 13 | 10
Not completed — Withdrawal by Subject | 10 | 6
Not completed — Not Selected | 0 | 1
Not completed — Continued treatment beyond 12 mo. | 58 | 50

BASELINE CHARACTERISTICS:
Groups:
- INTRON A (Interferon Alfa-2b): Interferon alfa-2b, recombinant for injection, 5 million international units (MIU)/m^2, administered daily by SC injection. Treatment was for a minimum of 6 months unless there was evidence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | INTRON A (Interferon Alfa-2b) | PEG Intron (Pegylated Interferon Alfa-2b) | Total
Number analyzed (Participants) | 173 | 171 | 344
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.6 (13.4) | 51.9 (12.8) | 51.7 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 75 | 142
  Male | 106 | 96 | 202

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cytogenetic Responses to PEG Intron and INTRON A at 12 Months
Description: Cytogenetic response (CR) was defined by the degree of suppression of Philadelphia chromosome (Ph^1) achieved during study treatment. For all participants continuing treatment after study conclusion, cytogenetic assessments were conducted locally as per standard of care. Determination of CR at 12 months were based on cytogenetic analysis of bone marrow aspirate samples. The CR criteria were based on the percentage (%) of PH^1-positive cells during study treatment. Protocol-defined CR criteria were Complete Response (0%), Partial Response (1-34%), Minor Response (35-90%), or No Response (>90%). Data for the analysis population was based on the intent-to-treat principle. Participants who were treatment failures at 6 months were considered cytogenetic non-responders. Recording of CR was independent of hematologic responses.
Time Frame: Up to 12 months
Population: All randomized participants analyzed on an intent-to-treat basis.
Measure: Count of Participants; unit: Participants
Arm/Group | INTRON A (Interferon Alfa-2b) | PEG Intron (Pegylated Interferon Alfa-2b)
Number analyzed (Participants) | 173 | 171
Participants
  Complete Response | 13 | 13
  Partial Response | 35 | 26
  Minor Respnse | 31 | 24
  No Respnse | 15 | 25
  Discontinued or No Hematologic CR at Month 6 | 78 | 83
  Participants with Missing Data | 1 | 0
Statistical Analysis 1: Comparison: INTRON A (Interferon Alfa-2b) vs PEG Intron (Pegylated Interferon Alfa-2b); Test type: Superiority or Other; p = 0.322, Fisher Exact — Analysis of Major Response; Missing data considered failures

2. Secondary Outcome: Number of Participants With Cytogenetic Response (CR) to PEG Intron and Intron A at 6 Months
Description: Cytogenetic response (CR) at 6 months, as at 12 months, was defined by the degree of suppression of Philadelphia chromosome (Ph^1) achieved during study treatment. The determination of CR at 6 months was based on cytogenetic analysis of bone marrow aspirate samples. The CR criteria were based on the percentage (%) of PH^1-positive cells during study treatment. Protocol-defined CR criteria were Complete (0%), Partial (1-34%), Minor (35-90%), or No Response (>90%). Data for the analysis population was based on the intent-to-treat principle. Participants who were treatment failures at 6 months were considered cytogenetic non-responders. Recording of CR was independent of hematologic responses.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of assigned treatment
Measure: Count of Participants; unit: Participants
Arm/Group | INTRON A (Interferon Alfa-2b) | PEG Intron (Pegylated Interferon Alfa-2b)
Number analyzed (Participants) | 173 | 171
Participants
  Complete Response: 0% Ph+ | 7 | 3
  Partial Response: 1-34% Ph+ | 19 | 23
  Minor Response: 35-90% Ph+ | 51 | 37
  No Response: >90% Ph+ | 48 | 61
  Participant with Missing Data | 48 | 47
Statistical Analysis 1: Comparison: INTRON A (Interferon Alfa-2b) vs PEG Intron (Pegylated Interferon Alfa-2b); Test type: Superiority or Other; p > 0.999, Fisher Exact — Analysis of Major Response; Missing data considered failures

3. Secondary Outcome: Number of Participants With Hematologic Responses to PEG Intron and Intron A at 6 Months
Description: Hematologic response at 6 months was assessed, while the hematologic response was measured at 3, 6, 9 and 12 months during the first year of study treatment. To be considered a hematologic responder a participant must have met all of the following criteria for a minimum of 28 days: WBC count <10,000/μL; platelet count <450,000/L; normal differential count in peripheral blood (manual differential count); no palpable spleen. Participants achieving a complete hematologic response at 3 months had the cytogenetic response evaluated at 3 months as well. Participants who achieved a complete hematologic response by 6 months continued treatment for another 6 months. Participants who failed to achieve a complete hematologic response after 6 months of treatment were considered treatment failures, and further treatment for this group was at the discretion of the treating physician. Participants may have continued to receive their assigned study medication for an additional 6 months.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of assigned treatment
Measure: Count of Participants; unit: Participants
Arm/Group | INTRON A (Interferon Alfa-2b) | PEG Intron (Pegylated Interferon Alfa-2b)
Number analyzed (Participants) | 173 | 171
Participants
  Complete Response | 98 | 91
  Treatment Failure | 44 | 52
  Missing | 31 | 28
Statistical Analysis 1: Comparison: INTRON A (Interferon Alfa-2b) vs PEG Intron (Pegylated Interferon Alfa-2b); Test type: Superiority or Other; p = 0.588, Fisher Exact — Analysis of Complete Response; Missing data considered failures

4. Secondary Outcome: Number of Participants With Overall Survival
Description: Participants were followed for survival; those who did not achieve a major cytogenetic response were discontinued from the study. For participants who completed 1 year of study treatment and continued to Year 2 and beyond, survival and disease progression every 3 months were assessed, and serious adverse events (SAEs) were reported. Participants were followed until resolution of any drug-related nonserious adverse event, and any SAE occurring while on the study or within 30 days of last dose of study drug. Participant death during survival follow-up was reported to the drug safety unit of the Sponsor. Each participant (whether discontinued or still on treatment) was followed every 3 months for survival and disease progression information. Overall survival was analyzed using the log-rank statistic, and the hazard ratio (HR) and 95% confidence interval (CI) for the HR were obtained using Cox's proportional hazards model.
Time Frame: Up to 2 years (24 months), and beyond
Population: All randomized participants who received at least one dose of assigned treatment
Measure: Count of Participants; unit: Participants
Arm/Group | INTRON A (Interferon Alfa-2b) | PEG Intron (Pegylated Interferon Alfa-2b)
Number analyzed (Participants) | 173 | 171
Participants
  Deaths | 15 | 17
  Survivors | 158 | 154
Statistical Analysis 1: Comparison: INTRON A (Interferon Alfa-2b) vs PEG Intron (Pegylated Interferon Alfa-2b); Test type: Superiority or Other; Cox Proportional Hazard = 0.859, 95% CI 2-sided [0.429 to 1.721] — Overall survival was analyzed using the log-rank statistic. The HR and 95% CI for the HR were obtained using Cox's proportional hazards model

ADVERSE EVENTS:
Time Frame: Up to One Year
Description: An AE is any physical or clinical change or disease experienced by the participant at any time during the course of the study, whether or not considered related to the use of the study drug. This includes the onset of new illness and the exacerbation of pre-existing conditions other than the indication under study. The population analyzed was all randomized participants who received at least one dose of study treatment. One randomized participant died before receiving treatment.
Groups:
- INTRON A, 5 MIU/m^2 Daily: Interferon alfa-2b, recombinant for injection, 5 million international units (MIU)/m^2, administered daily by SC injection. Treatment was for a minimum of 6 months (mo.) unless there was evidence of disease progression or unacceptable toxicity.
- PEG-Intron, 6.0 mcg/kg Weekly: Pegylated interferon alfa-2b, 6.0 microg/kg, administered weekly by subcutaneous (SC) injection. Treatment was for a minimum of 6 months unless there was evidence of disease progression or unacceptable toxicity.
Arm/Group | INTRON A, 5 MIU/m^2 Daily | PEG-Intron, 6.0 mcg/kg Weekly
All-Cause Mortality (participants affected / at risk) | 15/173 | 17/171
Serious Adverse Events (participants affected / at risk) | 62/173 | 74/171
Other Adverse Events (participants affected / at risk) | 170/173 | 168/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INTRON A, 5 MIU/m^2 Daily (N=173) | PEG-Intron, 6.0 mcg/kg Weekly (N=171)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HYPERGAMMAGLOBULINAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 0 (0)
CYANOSIS (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0)
TACHYARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 2 (2)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
OCULAR TOXICITY (Eye disorders) | 0 (0) | 1 (1)
VISUAL ACUITY REDUCED (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (3) | 3 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 2 (2)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
HIATUS HERNIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 2 (2) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 3 (4) | 6 (6)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 4 (5) | 3 (3)
ASTHENIA (General disorders) | 2 (4) | 2 (2)
CHEST PAIN (General disorders) | 3 (5) | 5 (5)
CHILLS (General disorders) | 2 (3) | 2 (2)
FATIGUE (General disorders) | 0 (0) | 3 (3)
HERNIA (General disorders) | 0 (0) | 1 (1)
HYPERTHERMIA (General disorders) | 1 (1) | 0 (0)
HYPOTHERMIA (General disorders) | 0 (0) | 1 (1)
MALAISE (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 6 (8) | 7 (8)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 2 (2) | 0 (0)
CYTOLYTIC HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATOMEGALY (Hepatobiliary disorders) | 0 (0) | 2 (2)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 1 (1)
JAUNDICE (Hepatobiliary disorders) | 1 (2) | 0 (0)
APPENDICITIS (Infections and infestations) | 2 (2) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
FUNGAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0)
INFECTED CYST (Infections and infestations) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 2 (2)
INJECTION SITE ABSCESS (Infections and infestations) | 2 (2) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 3 (3) | 2 (2)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
JOINT INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
ALANINE AMINOTRANSFERASE ABNORMAL (Investigations) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 2 (6)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 2 (5)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 0 (0) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 2 (3) | 2 (2)
HEPATITIS B VIRUS (Investigations) | 0 (0) | 1 (1)
LABORATORY TEST ABNORMAL (Investigations) | 1 (1) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 2 (2) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (1) | 2 (2)
ANOREXIA (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
CELL DEATH (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
BLAST CELL CRISIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
BLAST CRISIS IN MYELOGENOUS LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 1 (1)
COMA (Nervous system disorders) | 1 (1) | 0 (0)
CONVULSION (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (2) | 4 (5)
EPILEPSY (Nervous system disorders) | 0 (0) | 3 (3)
GRAND MAL CONVULSION (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 2 (2)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 2 (2)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
PARESIS (Nervous system disorders) | 1 (1) | 0 (0)
SCIATICA (Nervous system disorders) | 1 (1) | 2 (2)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0)
STATUS EPILEPTICUS (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 2 (2)
SYNCOPE VASOVAGAL (Nervous system disorders) | 2 (2) | 2 (2)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (2) | 1 (1)
DEPRESSION (Psychiatric disorders) | 3 (3) | 3 (3)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 2 (2)
CYSTOCELE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
METRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
AORTIC ANEURYSM (Vascular disorders) | 2 (2) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 2 (2)
VENA CAVA THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INTRON A, 5 MIU/m^2 Daily (N=173) | PEG-Intron, 6.0 mcg/kg Weekly (N=171)
ANAEMIA (Blood and lymphatic system disorders) | 8 (10) | 21 (43)
LEUKOPENIA (Blood and lymphatic system disorders) | 19 (32) | 19 (38)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 6 (7) | 13 (13)
NEUTROPENIA (Blood and lymphatic system disorders) | 9 (11) | 12 (29)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 35 (65) | 34 (74)
PALPITATIONS (Cardiac disorders) | 3 (3) | 10 (18)
EAR PAIN (Ear and labyrinth disorders) | 7 (63) | 10 (17)
TINNITUS (Ear and labyrinth disorders) | 6 (9) | 11 (17)
VERTIGO (Ear and labyrinth disorders) | 22 (36) | 23 (61)
CONJUNCTIVITIS (Eye disorders) | 6 (6) | 10 (15)
EYE PAIN (Eye disorders) | 12 (42) | 8 (25)
VISION BLURRED (Eye disorders) | 11 (14) | 13 (16)
ABDOMINAL PAIN (Gastrointestinal disorders) | 33 (59) | 39 (105)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 44 (108) | 51 (169)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 10 (15) | 7 (8)
CONSTIPATION (Gastrointestinal disorders) | 38 (130) | 36 (89)
DIARRHOEA (Gastrointestinal disorders) | 95 (314) | 104 (503)
DRY MOUTH (Gastrointestinal disorders) | 61 (157) | 57 (179)
DYSPEPSIA (Gastrointestinal disorders) | 23 (28) | 18 (33)
GASTRITIS (Gastrointestinal disorders) | 9 (14) | 3 (3)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 2 (2) | 10 (14)
NAUSEA (Gastrointestinal disorders) | 101 (429) | 111 (627)
ORAL PAIN (Gastrointestinal disorders) | 2 (3) | 12 (38)
STOMACH DISCOMFORT (Gastrointestinal disorders) | 16 (86) | 13 (51)
STOMATITIS (Gastrointestinal disorders) | 13 (16) | 9 (17)
TOOTHACHE (Gastrointestinal disorders) | 8 (11) | 9 (11)
VOMITING (Gastrointestinal disorders) | 53 (108) | 62 (178)
ASTHENIA (General disorders) | 81 (246) | 94 (400)
CHEST PAIN (General disorders) | 26 (68) | 26 (75)
CHILLS (General disorders) | 108 (254) | 115 (377)
FATIGUE (General disorders) | 105 (637) | 103 (929)
FEELING COLD (General disorders) | 9 (12) | 6 (24)
GAIT DISTURBANCE (General disorders) | 7 (7) | 12 (25)
INFLUENZA LIKE ILLNESS (General disorders) | 7 (10) | 10 (22)
INJECTION SITE ERYTHEMA (General disorders) | 17 (19) | 37 (80)
INJECTION SITE PAIN (General disorders) | 19 (31) | 20 (35)
INJECTION SITE RASH (General disorders) | 5 (7) | 11 (18)
INJECTION SITE REACTION (General disorders) | 6 (7) | 18 (48)
IRRITABILITY (General disorders) | 14 (34) | 9 (18)
MALAISE (General disorders) | 19 (45) | 27 (180)
OEDEMA PERIPHERAL (General disorders) | 11 (13) | 18 (28)
PAIN (General disorders) | 49 (135) | 48 (236)
PYREXIA (General disorders) | 133 (468) | 141 (1121)
THIRST (General disorders) | 4 (5) | 12 (16)
BRONCHITIS (Infections and infestations) | 13 (20) | 19 (25)
NASOPHARYNGITIS (Infections and infestations) | 18 (21) | 24 (56)
ORAL HERPES (Infections and infestations) | 5 (5) | 11 (17)
PHARYNGITIS (Infections and infestations) | 6 (9) | 10 (12)
RHINITIS (Infections and infestations) | 9 (9) | 9 (13)
SINUSITIS (Infections and infestations) | 10 (12) | 9 (17)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 (12) | 13 (17)
URINARY TRACT INFECTION (Infections and infestations) | 8 (10) | 15 (18)
PLATELET COUNT DECREASED (Investigations) | 11 (15) | 11 (19)
WEIGHT DECREASED (Investigations) | 69 (128) | 81 (122)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 11 (19) | 12 (39)
ANOREXIA (Metabolism and nutrition disorders) | 86 (218) | 103 (315)
DECREASED APPETITE (Metabolism and nutrition disorders) | 24 (52) | 29 (63)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 79 (401) | 87 (474)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 82 (337) | 80 (472)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 24 (93) | 48 (292)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 9 (30) | 7 (10)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 21 (54) | 14 (69)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 16 (25) | 17 (36)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 14 (34) | 16 (20)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 38 (89) | 33 (65)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 8 (14) | 16 (51)
MYALGIA (Musculoskeletal and connective tissue disorders) | 109 (416) | 99 (532)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 16 (28) | 17 (51)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 64 (304) | 56 (187)
AGEUSIA (Nervous system disorders) | 4 (5) | 10 (19)
AMNESIA (Nervous system disorders) | 10 (18) | 6 (10)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 12 (27) | 9 (15)
DIZZINESS (Nervous system disorders) | 68 (256) | 59 (252)
DYSGEUSIA (Nervous system disorders) | 34 (75) | 35 (101)
HEADACHE (Nervous system disorders) | 128 (716) | 132 (1362)
HYPOAESTHESIA (Nervous system disorders) | 14 (28) | 24 (43)
PARAESTHESIA (Nervous system disorders) | 17 (32) | 22 (34)
SCIATICA (Nervous system disorders) | 7 (10) | 10 (32)
SOMNOLENCE (Nervous system disorders) | 24 (44) | 20 (59)
TREMOR (Nervous system disorders) | 20 (44) | 23 (55)
ANXIETY (Psychiatric disorders) | 33 (61) | 42 (110)
DEPRESSED MOOD (Psychiatric disorders) | 3 (3) | 11 (22)
DEPRESSION (Psychiatric disorders) | 51 (111) | 58 (131)
INSOMNIA (Psychiatric disorders) | 57 (128) | 48 (150)
DYSURIA (Renal and urinary disorders) | 3 (4) | 10 (12)
COUGH (Respiratory, thoracic and mediastinal disorders) | 69 (122) | 56 (120)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 37 (98) | 38 (89)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 9 (14) | 3 (3)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 22 (37)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 11 (17) | 7 (13)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 36 (101) | 44 (109)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 19 (36) | 20 (30)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 20 (37)
ALOPECIA (Skin and subcutaneous tissue disorders) | 67 (84) | 53 (70)
DRY SKIN (Skin and subcutaneous tissue disorders) | 24 (48) | 18 (23)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 10 (14) | 11 (12)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 36 (55) | 42 (121)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 21 (49) | 30 (73)
PRURITUS (Skin and subcutaneous tissue disorders) | 37 (97) | 30 (57)
RASH (Skin and subcutaneous tissue disorders) | 27 (46) | 23 (56)
HYPOTENSION (Vascular disorders) | 9 (14) | 14 (20)

LIMITATIONS AND CAVEATS:
AE Preferred Terms were converted from WHO-ART dictionary to the MedDRA version 10.0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators have the right to publish or publicly present the results of the study. Principal Investigators further agree to provide to the Sponsor thirty (30) days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication. No publication or manuscript shall contain any trade secret information of the Sponsor or any proprietary or confidential information of the Sponsor.